CLINICAL TRIAL: NCT02939625
Title: Effects of Continuous and Bilevel Positive Airway Pressure During Exercise-induced Bronchoconstriction in Asthmatic Children: Controlled Clinical Trial, Randomized
Brief Title: NIV Application in the Treatment of Asthmatic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Daysi Tobelem, Md, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rehabilitation in asthma
Record Dates: First submitted 2016-10-12; First posted 2016-10-20 (Estimated); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Asthma; Child; Bronchial Spasm
MeSH Terms: conditions — Asthma; Bronchial Spasm | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- muscle training (Active Comparator): participants will breathing exercises for 20 min, then 40 min training with Threshold IMT therapy will be held in 7 sessions
  Interventions: Device: muscle training; Device: Continue Positive Airway Pressure; Device: bilevel positive airway pressure
- bilevel positive airway pressure (Active Comparator): participants will breathing exercises for 20 min, then 40 min bilevel (IPAP and EPAP 12 = 8 cm H2O), the therapy will be held in 7 sessions
  Interventions: Device: muscle training; Device: Continue Positive Airway Pressure; Device: bilevel positive airway pressure
- Continue Positive Airway Pressure (Active Comparator): participants will breathing exercises for 20 min, then 40 min CPAP (8 cm H2O) therapy will be held in 7 sessions
  Interventions: Device: muscle training; Device: Continue Positive Airway Pressure; Device: bilevel positive airway pressure

INTERVENTIONS:
Device: muscle training
Device: Continue Positive Airway Pressure
Device: bilevel positive airway pressure

SUMMARY:
Asthma is characterized by recurrent episodes of bronchospasm, bronchial hyperresponsiveness and chronic airway inflammation and pharmacological treatment for this condition is done with bronchodilators and anti-inflammatory.

DETAILED DESCRIPTION:
Pharmacologic therapy has clinical efficacy in the control, but the patient often does not adhere adequately.

There is need for further research into non-pharmacological therapies for clinical asthma control and in turn the use of CPAP and bilevel pressure in the airways has shown beneficial effects on autonomic modulation and bronchial responsiveness leading to the hypothesis that these therapies also have effects on the BIE.The aim of this study is to evaluate the effect of these non-pharmacological therapies in several variables and especially the BIE.

ELIGIBILITY:
Inclusion Criteria:

* Age between 5:11 years;
* Both sexes;
* Do not be included in any regular physical activity program;
* Having a diagnosis of asthma, according to the Global Initiative for Asthma (GINA);
* Not having received Theophylline or aminophylline and oral corticosteroids in the last 30 days;
* not have presented respiratory infection in the last two months;
* Signature of IC

Exclusion Criteria:

* Have done inhaled bronchodilator in less than 12 hours before the assessment;
* Inability to understand or perform any of the tests, due to physical and mental limitations;
* Intolerance proposed activities;
* Have heart disease inflammatory, congenital or ischemic origin;
* Being in the presence of any infectious process with fever.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2015-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Exhaled nitric oxide (part per billion) | 5 minutes
  assess the degree of inflammation of the respiratory system using expired fraction of nitric oxide before and after the different protocols applied

SECONDARY OUTCOMES:
Heart Rate Variability | 20 minutes
manovacuometry | 10 minutes
Pulmonary function test | 20 minutes
bioelectrical impedance | 10 minutes
Bronchoconstriction induced by stress | 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Maisi David Cabral, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] David MMC, Gomes ELFD, Mello MC, Costa D. Noninvasive ventilation and respiratory physical therapy reduce exercise-induced bronchospasm and pulmonary inflammation in children with asthma: randomized clinical trial. Ther Adv Respir Dis. 2018 Jan-Dec;12:1753466618777723. doi: 10.1177/1753466618777723. PMID 29865929